CLINICAL TRIAL: NCT06080321
Title: Oral Hygiene Compliance in Orthodontic Patients Using Active Reminders: A Randomized Controlled Clinical Trial
Brief Title: Oral Hygiene Compliance in Orthodontic Patients Using Active Reminders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: #9/2023
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Oral Hygiene; Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- WhatsApp messages (Experimental)
  Interventions: Other: WhatsApp reminders
- Instagram messages (Experimental)
  Interventions: Other: Instagram reminders
- Phone calls (Experimental)
  Interventions: Other: Phone calls
- App alerts (Active Comparator)
  Interventions: Other: Application alerts
- No active reminders (No Intervention)

INTERVENTIONS:
Other: WhatsApp reminders — Patients will receive active oral hygiene reminders in the form of WhatsApp messages one weekday each week. The standardized text message will be: "This is a message from the Orthodontic Clinic at Faculty of Dentistry, Alexandria reminding you that it is extremely important to brush your teeth for 2 minutes after every meal or at least 3 times daily. Cleaning your teeth will help to keep them healthy and beautiful."
  Arms: WhatsApp messages
Other: Instagram reminders — Patients will receive active oral hygiene reminders in the form of Instagram messages one weekday each week. The standardized text message will be: "This is a message from the Orthodontic Clinic at Faculty of Dentistry, Alexandria reminding you that it is extremely important to brush your teeth for 2 minutes after every meal or at least 3 times daily. Cleaning your teeth will help to keep them healthy and beautiful."
  Arms: Instagram messages
Other: Phone calls — Patients will receive active oral hygiene reminders in the form of phone calls one weekday each week. The structured phone call will be: "This is a message from the Orthodontic Clinic at Faculty of Dentistry, Alexandria reminding you that it is extremely important to brush your teeth for 2 minutes after every meal or at least 3 times daily. Cleaning your teeth will help to keep them healthy and beautiful."
  Arms: Phone calls
Other: Application alerts — Patients will download an app on their mobile phones which has cleaning tips, demonstrations and alerts. The structured message will be: "This is a message from the Orthodontic Clinic at Faculty of Dentistry, Alexandria reminding you that it is extremely important to brush your teeth for 2 minutes after every meal or at least 3 times daily. Cleaning your teeth will help to keep them healthy and beautiful."
  Arms: App alerts

SUMMARY:
The aim of the present study will be to determine if different forms of active reminders regarding oral hygiene compliance have an influence on the level of compliance within orthodontic patients

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a complete natural dentition.
* Patients who need to undergo orthodontic therapy using fixed appliances.
* Good oral hygiene, with no signs and symptoms of periodontal disease.
* Patients with no medical or mental problems.

Exclusion Criteria:

* Patients with health risks associated with periodontal probing.
* Syndromic patients ex; Down syndrome.
* Previous orthodontic treatment.
* Patients with carious teeth

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Gingival bleeding | up to 6 months
  This will be assessed using the bleeding index (BI) upon probing the mesio-buccal, direct buccal, and disto-buccal aspects of the gingival sulci of the teeth. BI scoring ranges from 0-2; 0: no bleeding after 30 seconds, 1: bleeding after 30 seconds, 2: immediate bleeding
Gingival inflammation | up to 6 months
  This will be assessed using the modified gingival index (MGI). One MGI measurement of the buccal marginal gingiva for each tooth will be scored. Scoring ranges from 0-4 where 0 indicates absence of inflammation, 1: mild inflammation (marginal or papillary unit), 2: mild inflammation (entire marginal and papillary unit), 3: moderate inflammation, and 4: severe inflammation
Plaque accumulation | up to 6 months
  This will be assessed using the plaque index (PI). One PI measurement will be recorded for the buccal surface of each tooth. Scoring ranges from 0-5; where 0 indicates absence of plaque, 1: discontinuous plaque band at gingival margin, 2: up to 1 mm continuous plaque band at gingival margin, 3: plaque band wider than 1 mm but less than 1/3 of the surface, 4: plaque band between 1/3 and 2/3 of the surface, and 5: plaque covering 2/3 or more of the surface
Visual examination of white spot lesions | up to 6 months
  The presence of white spot lesions located on the buccal surface gingival to the archwire will be examined visually on the maxillary and mandibular six anterior teeth after being air dried for 5 seconds. Scoring ranges from 0-3; where 0: no visible white spot or surface disruption, 1: visible white spot without surface disruption, 2: visible white spot with roughened surface, 3: visible white spot requiring restoration.

CONTACTS AND LOCATIONS:
Overall Officials: Samar M Adel, PhD, Principal Investigator — Alexandria University; Nikhilesh R Vaid, PhD, Study Chair — Department of Orthodontics, Saveetha Dental College, Saveetha Institute of Medical and Technical Sciences, Chennai, India; Eiman Marzouk, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt